CLINICAL TRIAL: NCT02178644
Title: Pilot Trial of KD018 With Neo-Adjuvant Concurrent Chemo-Radiation Therapy in Patients With Locally Advanced Rectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1404013708
Record Dates: First submitted 2014-06-26; First posted 2014-07-01 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Drug Therapy; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemo with concomitant Capecitabine and KD018 (Experimental): Patients will receive a course of chemo-radiation with concomitant Capecitabine and KD018, and to compare this to the toxicity seen in patients treated with Capecitabine and radiation therapy alone, in patients with T3-T4 and N0-N2, M0 rectal cancer.
  Interventions: Drug: Chemo with concomitant Capecitabine and KD018

INTERVENTIONS:
Drug: Chemo with concomitant Capecitabine and KD018 — Patients will receive a course of chemo-radiation with concomitant Capecitabine and KD018, and to compare this to the toxicity seen in patients treated with Capecitabine and radiation therapy alone, in patients with T3-T4 and N0-N2, M0 rectal cancer.
  Other Names: KD018; Capecitabine; Neo-Adjuvant Concurrent Chemo-Radiation Therapy

SUMMARY:
This pilot study focuses on KD018 and will investigate the effect of this agent on reducing the Gastrointestinal (GI) toxicity associated with combined modality therapy of locally-advanced rectal cancer.

DETAILED DESCRIPTION:
This pilot study focuses on KD018, a standardized and well-characterized Chinese herbal medicine, and will investigate the effect of this agent on reducing the GI toxicity associated with combined modality therapy of locally-advanced rectal cancer. In this study, KD018 will be administered concomitantly with Capecitabine and pelvic radiation therapy (RT) in the neoadjuvant setting, with the hypothesis that KD018 will reduce the gastrointestinal side effects, namely diarrhea, secondary to treatment with Capecitabine plus external beam radiation therapy (EBRT).

The primary endpoint of the study is to investigate the grade 3-4 toxicity rate associated with a course of chemo-radiation with concomitant Capecitabine and KD018, and to compare this to the toxicity seen in patients treated with Capecitabine and radiation therapy alone, in patients with T3-T4 and N0-N2, M0 rectal cancer. Secondary objectives include the assessment of radiographic response to therapy (using pelvic MRI) and assessment of the pathologic CR rate by examination of the pathologic specimen. In addition, we will perform an analysis of plasma levels of pro-inflammatory cytokines and chemokines.

This trial is designed to accrue approximately 24 patients over the course of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed T3-T4 and N0-N2, M0 adenocarcinoma of the rectum with the inferior margin within 16 cm from the anal verge.
* Patients must have had a Transrectal ultrasound (TRUS)/endoscopic ultrasound (TEUS) staging within two months prior to treatment start.
* Patients must have had a pelvic MRI within 28 days prior to the initiation of treatment.
* Patient must have the ability to swallow multiple capsules.
* Women of child bearing potential between the ages of 18 and 60 years of age must have a negative urine pregnancy test prior to undergoing simulation in preparation for radiation therapy to the pelvis.
* ECOG performance status of 0 to 1 within 28 days prior to initiation of treatment.
* Patients must have normal organ and marrow function as defined below. All laboratory values must be obtained within 14 days prior to initiation of treatment:
* absolute neutrophil count >= 1,500/mcL
* platelets >= 100,000/mcL
* hemoglobin >= 8.0 g/ dL
* serum bilirubin < 1.5 times the upper limit of of normal (ULN)
* serum AST, ALT < 2.5 times ULN
* serum Creatinine ≤ 1.5 times ULN
* The effects of radiation on the developing human fetus are known to be teratogenic. For this reason, all women and sexually active men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

* History of clinically significant Crohn's disease or inflammatory bowel disease (IBD).
* Active collagen vascular disease.
* History of previous abdominal or pelvic radiation therapy.
* History of previous systemic chemotherapy unless given curatively for other malignancy now > 5 years without evidence of recurrence.
* Patients with suspected or confirmed poor compliance, mental instability, or prior or current alcohol or drug abuse deemed by the investigator to be likely to affect their ability to sign the informed consent, or undergo study procedures will be excluded.
* Pregnant women are excluded from this study because radiation has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with either KD018 or Capecitabine, breastfeeding should be discontinued if the mother is treated.
* Patients with known HIV infection or viral hepatitis.
* Patients with Dihydropyrimidine dehydrogenase (DPD) deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-07; Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Grade 3-4 Toxicity Rate | Up to 10 Months
  Grade 3-4 toxicity rate will be described as greatest toxicity per patient/total patients evaluable for toxicity +/- 95% confidence interval.
pCR Rate | Up to 10 Months
  pCR (CR = Complete Response) rate will be defined as number of patients with pathologic complete response divided by number of patients treated (pCR IIT) and divided by those undergoing surgical resection (pCR actual) +/- 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Susan A Higgins, M.D., M.S., Principal Investigator — Yale University
Locations (1):
- Yale Cancer Center, New Haven, Connecticut, United States